CLINICAL TRIAL: NCT03758365
Title: A Randomized, Evaluator Blinded, Within Subject, Single-Centre Evaluation of the Vasoconstriction Properties of MC2-01 Cream, Compared to 5 Other Corticosteroids in Healthy Subjects
Brief Title: Evaluation of the Vasoconstriction Properties of MC2-01 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MC2-01-C4
Record Dates: First submitted 2018-11-13; First posted 2018-11-29 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Vasoconstriction
MeSH Terms: interventions — calcipotriene; Clobetasol; betamethasone-17,21-dipropionate; Triamcinolone Acetonide; hydrocortisone-17-butyrate; Desonide

STUDY DESIGN:
Intervention Model Description: Single application, intra individual comparison on mini-test sites (n=7)
Who Masked: Outcomes Assessor
Masking Description: Visual assessments of potential skin blanching will be made independently by 2 trained observers, according to a grading scale (0 to 4)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- MC2-01 Cream (Experimental): Single application of MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream
  Interventions: Drug: MC2-01 Cream
- Clobetasol propionate 0.05% lotion (Active Comparator): Single application of Clobetasol propionate 0.05%,
  Interventions: Drug: Clobetasol Propionate 0.05% Lotion
- Betamethasone dipropionate 0.05% cream (Active Comparator): Single application of Betamethasone dipropionate 0.05%,
  Interventions: Drug: Betamethasone Dipropionate 0.05% Cream
- Triamcinolone acetonide 0.1% cream (Active Comparator): Single application of Triamcinolone acetonide 0.1%,
  Interventions: Drug: Triamcinolone Acetonide 0.1% Cream
- Hydrocortisone Butyrate 0.1% cream (Active Comparator): Single application of Hydrocortisone Butyrate 0.1% Cream
  Interventions: Drug: Hydrocortisone Butyrate 0.1% Cream
- Desonide 0.05% cream (Active Comparator): Single application of Desonide 0.05%
  Interventions: Drug: Desonide 0.05% Cream
- Vehicle cream (Placebo Comparator): Single application of Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: MC2-01 Cream — Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
  Other Names: Calcipotriol + Betamethasone dipropionate cream
  Arms: MC2-01 Cream
Drug: Clobetasol Propionate 0.05% Lotion — Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
  Other Names: Clobex
  Arms: Clobetasol propionate 0.05% lotion
Drug: Betamethasone Dipropionate 0.05% Cream — Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
  Other Names: Betamethasone Dipropionate
  Arms: Betamethasone dipropionate 0.05% cream
Drug: Triamcinolone Acetonide 0.1% Cream — Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
  Other Names: Triamcinolone acetonide
  Arms: Triamcinolone acetonide 0.1% cream
Drug: Hydrocortisone Butyrate 0.1% Cream — Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
  Other Names: Locoid® cream
  Arms: Hydrocortisone Butyrate 0.1% cream
Drug: Desonide 0.05% Cream — Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
  Other Names: Desowen® cream
  Arms: Desonide 0.05% cream
Drug: Vehicle — Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
  Other Names: Vehicle cream
  Arms: Vehicle cream

SUMMARY:
The objective of this trial is to compare the vasoconstriction potential

DETAILED DESCRIPTION:
The objective of this trial is to compare the vasoconstriction potential (skin blanching effect) of MC2-01 cream with 5 comparators and MC2-01 vehicle using the human skin blanching test (McKenzie-Stoughton's test).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years to 50 years old having signed and dated an informed consent,
2. Non-smoker subjects,
3. Subjects demonstrating adequate vasoconstriction to Diprolene® cream within 15 days prior to dosing (unoccluded application of Diprolene® cream for 4-6 hours must show a visual score of skin blanching of at least one unit (visual scale (0-4)),
4. Subjects without signs of skin irritation/disease/disorders/symptoms or blemishes on test sites (e.g. erythema, dryness, roughness, scaling, scars, moles, sunburn),
5. Female subjects of non-childbearing potential defined as surgically sterile or post-menopausal (at least one year post cessation of menses),
6. Female subjects of childbearing potential who have been, in the opinion of the Investigator, using an approved method of birth control (e.g. oral contraception pill or patch, intra-uterine devices, contraceptive implants or vaginal rings, condoms, bilateral tubal ligation) at trial entry and agree to continue until the end of the last trial visit,
7. Female subjects of childbearing potential must have a negative urine pregnancy test at screening visit and at Day 1 to continue,
8. Subjects willing and able to follow all the trial procedures and complete the whole trial,
9. Subjects affiliated to a social security system.

Exclusion Criteria:

1. Female subjects who are breastfeeding,
2. Use of topical corticosteroids on the test areas (forearms) within 4 weeks prior to the screening phase,
3. Use of systemic drugs which may interfere with the blanching reaction including, but not limited to, corticosteroids and other vasoactive drugs (nitrates derivatives, antihypertensive, phenylpropanolamine, diphenhydramine, pseudo-ephedrine, antihistamines, non-steroidal anti-inflammatory drug and aspirin/acetylsalicylic acid), within two weeks prior to screening visit,
4. Use of any other medication would interfere with the trial results, in particular topical drugs applied on the test area within two weeks prior to screening visit,
5. Subjects having a caffeine (i.e. coffee, cola, soft-drinks containing caffeine) intake greater than 500mg per day (1 cup of coffee contains approximately 85mg of caffeine) within one day prior to screening visit and until the end of the last visit of the test phase,
6. Subjects with a history of drug or alcohol abuse/addiction.
7. Abnormal pigmentation of the skin or skin type, that could, in any way, confound interpretation of the trail results (skin type V to VI on the Fitzpatrick scale),
8. Subjects with obvious difference in skin color between arms,
9. Subjects with any of the following conditions present on the test areas: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, atrophic skin, and striae atrophicae, fragility of skin veins, ichthyosis and ulcers,
10. Any current systemic or cutaneous disease that could in any way confound interpretation of the trial results (e.g. atopic dermatitis, contact eczema, or psoriasis),
11. Known or suspected hypersensitivity to any component(s) of Investigational Medical Product (IMP),
12. Subjects with current participation in any other interventional clinical, based on interview of the subject,
13. Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within the last 4 weeks prior to screening phase,
14. Previously enrolled in this clinical trial,
15. Subjects who do not accept to avoid strenuous physical activity nor alcohol intake during the study.
16. In the opinion of the (sub)investigator, subjects who are unlikely to comply with the Clinical Trial Protocol (e.g. alcoholism, drug dependency or psychotic state),
17. Subjects in close affiliation with the trial personnel (e.g. immediate family member or subordinate), subjects being a member of the clinical trial personnel, or being an employee of the sponsor or a Contract Research Organisation (CRO involved in the trial,
18. Subjects impossible to contact in case of emergency,
19. Subjects who are in an exclusion period in the National Biomedical Research Register of the French Ministry of Health at randomization,
20. Subjects under guardianship, hospitalized in a public or private institution, for a reason other than the research or subject deprived of freedom.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine QUEILLE-ROUSSEL, MD, Principal Investigator — CPCAD, Centre de Pharmacologie Clinique Appliquée à la Dermatologie
Locations (1):
- CPCAD, Nice, France

IPD SHARING:
Plan to Share IPD: No
Single site study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 07-Nov-2018. Last Subject Last Visit: 23-Nov-2018
Pre-assignment Details: The study consist of a screening period up to 15 day prior to randomization, a test period and a follow-up period.
  The study design is a within subject evaluation of the vasoconstriction properties of MC2-01 cream compared with vehicle cream and 5 other corticosteroids. All subjects received therefore a single treatment with all 7 products.
Groups:
- MC2-01 Cream + Comparators: Single application of 7 different treatments, where different sections on the arm was randomized to the following interventions:
  1. - MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream
  2. - Clobetasol Propionate 0.05% Lotion
  3. - Betamethasone Dipropionate 0.05% Cream
  4. - Triamcinolone Acetonide 0.1% Cream
  5. - Hydrocortisone Butyrate 0.1% Cream
  6. - Desonide 0.05% Cream
  7. - Vehicle Cream
  to perform visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
Period: Overall Study
Arm/Group | MC2-01 Cream + Comparators
Started | 36
MC2-01 Cream | 36
Clobetasol Propionate 0.05% Lotion | 36
Betamethasone Dipropionate 0.05% Cream | 36
Triamcinolone Acetonide 0,1% Cream | 36
Hydrocortisone Butyrate 0.1% Cream | 36
Desonide 0.05% Cream | 36
Vehicle Cream | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients received all 7 types of treatments.
Arm/Group | MC2-01 Cream + Comparators
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 36 patients participated and they received all types of treatment. Therefore analyses of the 7 treatments arms were done for all 36 patients.
  years | 34.36 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 36
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I | 0
  II | 9
  III | 24
  IV | 3
  V | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Vasoconstriction Potential (Skin Blanching Effect) of the MC2-01 Cream With Active Comparators and Vehicle
Description: Blanching of the skin will be assessed individually by two trained observers blinded to treatment. The observers will score the blanching of the skin from 0-4 (0 = No change in color skin; 1 = Slight (barely visible) blanching; 3 = Obvious blanching; 4 = Blanching judged to be maximal). The results is presented as Mean ± SD.
Time Frame: Day 2
Population: As the study design is a within subject evaluation of the vasoconstriction properties of MC2-01 cream compared with vehicle cream and 5 other corticosteroids, all 36 enrolled subjects received a single treatment with all 7 products.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MC2-01 Cream + Comparators: Single application of MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream
  MC2-01 Cream: Single application, visual evaluation of skin blanching and local tolerability, physical examination and safety evaluation
Arm/Group | MC2-01 Cream + Comparators
Number analyzed (Participants) | 36
score on a scale
  MC2-01 Cream | 1.66 (0.57)
  Clobetasol Propionate 0.05% Lotion | 3.05 (0.65)
  Betamethasone Dipropionate 0.05% Cream | 2.45 (0.61)
  Triamcinolone Acetonide 0.1% Cream | 1.92 (0.89)
  Hydrocortisone Butyrate 0.1% Cream | 2.06 (0.70)
  Desonide 0.05% Cream | 2.11 (0.85)
  Vehicle Cream | 0.14 (0.25)

2. Primary Outcome: Compare Local Tolerability of the MC2-01 Cream With Active Comparators and Vehicle
Description: The local tolerability of the creams will be assesed using a predefined scale: 0 = No reaction; 0.5 = Only slight erythema; 1 = Only erythema; 2 = Erythema with papules or oedema; 3 = Erythema, oedema with papules, oedema with vesicle; 4 = Blisters
Time Frame: Day 2
Population: The local tolerance score is presented as number of participants with observed local reaction by trial product and severity.
Measure: Count of Participants; unit: Participants
Groups:
- MC2-01 Cream + Comparators: Single application of 7 different treatments, where different sections on the arm was randomized to the following interventions:
  1. - MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream
  2. - Clobetasol Propionate 0.05% Lotion
  3. - Betamethasone Dipropionate 0.05% Cream
  4. - Triamcinolone Acetonide 0.1% Cream
  5. - Hydrocortisone Butyrate 0.1% Cream
  6. - Desonide 0.05% Cream
  7. - Vehicle Cream
  to perform visual evaluation of local tolerability, physical examination and safety evaluation
Arm/Group | MC2-01 Cream + Comparators
Number analyzed (Participants) | 36
Participants
  MC2-01 Cream: No reaction | 36
  MC2-01 Cream: Only Slight reaction | 0
  MC2-01 Cream: Only erythema | 0
  MC2-01 Cream: Erythema with papules or oedema | 0
  MC2-01 Cream: Erythema, oedema with papules, oedema with vesicle | 0
  MC2-01 Cream: Blisters | 0
  Clobetasol Propionate 0.05% Lotion: No reaction | 36
  Clobetasol Propionate 0.05% Lotion: Only Slight reaction | 0
  Clobetasol Propionate 0.05% Lotion: Only erythema | 0
  Clobetasol Propionate 0.05% Lotion: Erythema with papules or oedema | 0
  Clobetasol Propionate 0.05% Lotion: Erythema, oedema with papules, oedema with vesicle | 0
  Clobetasol Propionate 0.05% Lotion: Blisters | 0
  Betamethasone Dipropionate 0.05% Cream: No reaction | 36
  Betamethasone Dipropionate 0.05% Cream: Only Slight reaction | 0
  Betamethasone Dipropionate 0.05% Cream: Only erythema | 0
  Betamethasone Dipropionate 0.05% Cream: Erythema with papules or oedema | 0
  Betamethasone Dipropionate 0.05% Cream: Erythema, oedema with papules, oedema with vesicle | 0
  Betamethasone Dipropionate 0.05% Cream: Blisters | 0
  Triamcinolone Acetonide 0.1% Cream: No reaction | 36
  Triamcinolone Acetonide 0.1% Cream: Only Slight reaction | 0
  Triamcinolone Acetonide 0.1% Cream: Only erythema | 0
  Triamcinolone Acetonide 0.1% Cream: Erythema with papules or oedema | 0
  Triamcinolone Acetonide 0.1% Cream: Erythema, oedema with papules, oedema with vesicle | 0
  Triamcinolone Acetonide 0.1% Cream: Blisters | 0
  Hydrocortisone Butyrate 0.1% Cream: No reaction | 36
  Hydrocortisone Butyrate 0.1% Cream: Only Slight reaction | 0
  Hydrocortisone Butyrate 0.1% Cream: Only erythema | 0
  Hydrocortisone Butyrate 0.1% Cream: Erythema with papules or oedema | 0
  Hydrocortisone Butyrate 0.1% Cream: Erythema, oedema with papules, oedema with vesicle | 0
  Hydrocortisone Butyrate 0.1% Cream: Blisters | 0
  Desonide 0.05% Cream: No reaction | 36
  Desonide 0.05% Cream: Only Slight reaction | 0
  Desonide 0.05% Cream: Only erythema | 0
  Desonide 0.05% Cream: Erythema with papules or oedema | 0
  Desonide 0.05% Cream: Erythema, oedema with papules, oedema with vesicle | 0
  Desonide 0.05% Cream: Blisters | 0
  Vehicle Cream: No reaction | 36
  Vehicle Cream: Only Slight reaction | 0
  Vehicle Cream: Only erythema | 0
  Vehicle Cream: Erythema with papules or oedema | 0
  Vehicle Cream: Erythema, oedema with papules, oedema with vesicle | 0
  Vehicle Cream: Blisters | 0

ADVERSE EVENTS:
Time Frame: AEs were collected/assessed from the time the informed consent form was signed at the screening visit, which could occur up to 14 days prior to the test period, during the 2 day's test period and until the follow-up visit, 15 days following the test period, had occurred. AEs assessed as reasonably possibly related to the trial medication had to be followed until they were resolved or until the medical condition of the subject was stable.
Description: 36 patients participated in the study and all patients received all 7 types of treatments. Therefore data for the 'All-Cause Mortality', 'Serious Adverse Events' and 'Other Adverse Events' fields are included and assessed for all types of medication.
Arm/Group | MC2-01 Cream | Clobetasol Propionate 0.05% Lotion | Betamethasone Dipropionate 0.05% Cream | Triamcinolone Acetonide 0.1% Cream | Hydrocortisone Butyrate 0.1% Cream | Desonide 0.05% Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The final report, the protocol and the raw date are the exclusive property of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT03758365/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT03758365/SAP_001.pdf